CLINICAL TRIAL: NCT05323942
Title: The Effect of Sleep Hygiene and Exercise Therapy on Bruxism, Sleep Habits, and Oral Habits in Children With Sleep Bruxism.
Brief Title: The Effect of Sleep Hygiene and Exercise Therapy in Children With Sleep Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aysenur Tuncer, Assistant Professor, Faculty, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/92
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-06

CONDITIONS: Sleep Bruxism, Childhood
Keywords: Bruxism; Sleep Habits; Oral Habits; Children
MeSH Terms: conditions — Sleep Bruxism; Bruxism | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education and Exercise Therapy Group (Other): Children and their parents were trained about bruxism, parafunctional oral habits, and sleep hygiene education. Therapeutic exercises about head-neck posture, breathing, and relaxation were given for 8 weeks.
  Interventions: Other: Education and Exercise Therapy Group

INTERVENTIONS:
Other: Education and Exercise Therapy Group — 82 children were evaluated. Among those, 37 volunteered children were trained and demonstrated in practice about bruxism, parafunctional oral habits, sleep hygiene education, and 5x5 therapeutic exercises. Therapeutic exercises program 5x5 included breathing exercises, head-neck, and scapular posture exercises which included jaw muscle and neck muscle stretching and strengthening exercises. They were asked to repeat each exercise with 5 set and 5 times a day for 8 weeks.
  Sleep hygiene education was given to parents and children with explanation of the parafunctional oral habits to raise awareness about being conscious about the oral habits. Sleep hygiene education includes routines about bedtime, sleeping room environment, and timing for exercise.

SUMMARY:
The aims of this study were to determine the relationship between sleep bruxism, oral habits, and sleep habits and establish treatment approaches in children.

DETAILED DESCRIPTION:
This cross-sectional study was conducted on children aged between 6-and 13 years, diagnosed with sleep bruxism (SB). Initially, 82 children with a diagnosis of SB were evaluated. Among those, 37 children volunteered were followed for 8 weeks to investigate the effects of the education, sleep hygiene and therapeutic exercise program.

Sleep hygiene education includes routines about bedtime, sleeping room environment, and timing for exercise.

Therapeutic exercises program 5x5 included breathing exercises, head-neck, and scapular posture exercises which included jaw muscle and neck muscle stretching and strengthening exercises. They were asked to repeat each exercise 5 times and 5 times a day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 - 13,
* Having a diagnosis of sleep bruxism,,
* And a parent signing informed consent for participation in the study.

Exclusion Criteria:

* Children who received orthodontic treatment,
* Children with the dentofacial anomaly, a history of TMJ surgery, having a medical history of neurological or psychiatric disease
* and those who could not cooperate were excluded from the study.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2020-03-08 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at 8 weeks | Baseline, 8 weeks
  The pain was measured with the Visual Analogue Scale (VAS) and the degree of pain was questioned in various situations. The children were told to mark the value of 0 when they felt no pain, 10 when they felt excruciating pain, and to mark the pain they felt within this range. And it was supported by facial expressions.
  Headache when waking up in the morning, jaw pain when waking up in the morning, jaw pain while eating, jaw pain after meals, and jaw pain before going to bed at night were questioned and each was measured by VAS.
Change from Baseline in Children's Sleep Habits Questionnaire (CSHQ) at 8 weeks | Baseline, 8 weeks
  Children's Sleep Habits Questionnaire (CSHQ) investigate children's sleep habits and sleep-related problems, and its Turkish validity and reliability were used. After giving the necessary information about the questionnaire to the parents, they were asked to fill it out.
  The CSHQ has satisfactory psychometric properties in children and has been used in the investigation of sleep in children. The form consists of 33 items in total. There are eight subscales in the scale, which can be listed as bedtime resistance, delayed falling asleep, sleep duration, sleep anxiety, night awakenings, parasomnias, impaired breathing during sleep, and daytime sleepiness.
Change from Baseline in Oral Habits at 8 weeks | Baseline, 8 weeks
  The evaluation was made with the 21-item Oral Habits Questionnaire (OAA). Each item was evaluated according to the frequency of complaints as "4 = always; 3 = most of the time; 2 = sometimes; filled with 1 = several times or 0 = none".
  A person's overall score can range from 0 to 84. A low overall score indicates positive oral habit, while a higher score indicates negative oral habit.
  After making sure that the questions were correctly understood by the children, the markings of the answers were made by the practitioner.

SECONDARY OUTCOMES:
Change from Baseline in Temporomandibular Joint (TMJ) Range of Motion (ROM) at 8 weeks | Baseline, 8 weeks
  TMJ ROM was analyzed as active and passive. Maximal mouth opening and right-left shifts were measured using a linear ruler. Active and passive maximal mouth opening, right and left lateral displacement, and protrusion of the TMJ were measured in millimeters (mm) based on reference points in the maxillary and mandibular anterior incisors.
  Crepitation and joint clicking sounds were questioned during mouth opening and closing, and normal line deviations were detected during mouth opening.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No